CLINICAL TRIAL: NCT01327118
Title: Headache Inducing Characteristics and Possible Changes in Cerebral Blood Flow After Administration of Prostaglandin F2alpha
Brief Title: Prostaglandin F2alpha in a Human Headache Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Danish Headache Center, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: DHC-PGF2-2010
Record Dates: First submitted 2011-03-29; First posted 2011-04-01 (Estimated); Last update posted 2011-04-14 (Estimated); Status verified 2010-07

CONDITIONS: Headache
MeSH Terms: conditions — Headache | interventions — Dinoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoton sodium chloride (Placebo Comparator)
  Interventions: Drug: Isoton sodium chloride
- Prostaglandin F2alpha (Active Comparator)
  Interventions: Drug: Prostaglandin F2alpha

INTERVENTIONS:
Drug: Prostaglandin F2alpha — intravenous injection
  Other Names: Dinoprost
  Arms: Prostaglandin F2alpha
Drug: Isoton sodium chloride — intravenous injection
  Other Names: placebo
  Arms: Isoton sodium chloride

SUMMARY:
The hypothesis of this study is that PGF2alpha does not induce headache or dilatation of brain vessels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Primary Headache
* Headache on the day of the investigation
* Hypertension
* Hypotension
* Pregnant/nursing
* Daily intake of medication (except oral contraceptives)
* Cardiovascular or central nervous system (CNS) disease
* Drug/alcohol abuse
* Psychiatric disease

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Headache score on a 10-point verbal rating scale (VRS) 0 indicated no headache; 1 indicated a different sensation, pounding or throbbing, but not necessarily painful; 5 indicated moderate headache and 10 indicated worst imaginable headache | 24 h.
  incidence of headache

SECONDARY OUTCOMES:
Blood flow velocity in the middle cerebral artery (VMCA) measured by a Transcranial Doppler (TCD) ultrasonography (2MHz) | in-hospital 2 h.
  changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
diameter of superficial temporal artery and radial artery measured by a high resolution ultrasound scanner, C-scan | in-hospital 2 h.
  changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
mean arterial blood pressure (MAP), heart rate (HR), end-tidal partial pressure of pCO2 (PetCO2), transcutaneous arterial oxygen saturation (SAT) measured by ProPac Encore® | in-hospital 2 h.
  changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.
electrocardiography (ECG) | in-hospital 2 h.
  changes from base line recorded every 10th min. until time 90 min on day 1 and day 2. The infusion takes 25 min from time 0.

CONTACTS AND LOCATIONS:
Overall Officials: Troels Wienecke, MD,PhD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark